CLINICAL TRIAL: NCT05854693
Title: Exploring the Effect of Trans-cranial Direct Current Stimulation on Craving and Serum BDNF of Patients With Alcohol Dependence
Brief Title: Trans-cranial Direct Current Stimulation on Alcohol Craving
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCHIRB-10907010
Record Dates: First submitted 2023-04-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2022-05

CONDITIONS: Alcohol Dependence
Keywords: Transcranial Direct Current Stimulation, craving
MeSH Terms: conditions — Alcoholism | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Experimental): The intervention consisted of 10 daily 20-min sessions of bilateral prefrontal tDCS (anodal-right/cathodal-left, 2mA; 1 × 1 Mini-CT)
  Interventions: Device: transCranial direct current stimulation
- Sham tDCS (Sham Comparator): The sham group consisted of 10 daily 20-min sessions of sham stimulation
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: transCranial direct current stimulation — The intervention consisted of 20 daily 20-min sessions of bilateral prefrontal tDCS
  Arms: Active tDCS
Device: sham stimulation — The sham group consisted of 10 daily 20-min sessions of sham stimulation
  Arms: Sham tDCS

SUMMARY:
The goal of thisclinical trial is to investigate the efficacy of trans cranial direct current stimulation (tDCS) for alcohol craving in individuals with alcohol dependence. The main question it aims to answer is whether 10 sessions of tDCS can reduce craving for alcohol.

Participants will be randomized into active group and sham group. Researchers will compare the severity of craving in these groups.

DETAILED DESCRIPTION:
Craving is defined as strong desire for substance use, and is one of the core symptoms of alcohol dependence which is highly correlated with relapse. Transcranial direct current stimulation (tDCS) involves applying a small direct current (1-2mA) to the prefrontal cortex; its therapeutic effect for depression and cognition has been demonstrated by several randomized studies. Our preliminary study has shown that tDCS has the potential to reduce craving in alcohol-dependent patients without adverse events. Furthermore, our previous studies have shown that serum brain-derived neurotrophic factor (BDNF) level is elevated after alcohol withdrawal. The current study aims at examining the association between craving and serum BDNF level in alcohol-dependent patients receiving tDCS. The study recruits 40 patients with alcohol dependence. Patients will receive tDCS for 2 weeks during admission, and followed for 2 weeks after tDCS. We'll compare their improvements in craving scores every week, and investigate the correlation between craving and serum BDNF level. This study will bring innovations to the treatment of alcohol dependence based on our previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 20-65 years of age
2. have sufficient cognitive function to understand the study and complete the informed consent process
3. Be diagnosed with alcohol dependence as defined by DSM-IV through a structured interview (Mini-International Neuropsychiatric Interview, M.I.N.I.)

Exclusion Criteria:

1. Intellectual disabilities
2. bipolar disorder
3. Psychosis (schizophrenia)
4. Major physical illness (brain hemorrhage, brain tumor, myocardial infarction, epilepsy or history of seizures)
5. intracorporeal electronic or metal implants (e.g., cardiac pacemaker)
6. Pregnant or breastfeeding women
7. Allergy to headgear and electrode materials
8. Trauma or infection to the head
9. Intracranial space occupied lesion (such as brain tumor, AVM, etc.) or patients who have undergone brain surgery, meningitis and encephalitis
10. Patients who are expected to undergo brain and major surgery during the trial period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol craving | Before intervention (week 0) and after intervention (week 2)
  Measured by visual analog scale, from 0-10

SECONDARY OUTCOMES:
Change in brain-derived neurotrophic factor (BDNF) | Before intervention (week 0) and after intervention (week 2)
  Serum level of BDNF

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei City Hospital, Taipei, Taipei CITY, Taiwan

IPD SHARING:
Plan to Share IPD: No